CLINICAL TRIAL: NCT07120126
Title: Evaluation of the Effect of Sonic Activation Using the EDDY Device on Root Canal Microbiota and Postoperative Pain in Teeth With Asymptomatic Apical Periodontitis: A Prospective Randomized Controlled Clinical Trial
Brief Title: Effect of EDDY Sonic Irrigation on Root Canal Microbiota and Pain in Asymptomatic Apical Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abdulkadir Tiftik,DDS (Other)
Responsible Party: Sponsor-Investigator, Abdulkadir Tiftik,DDS, Specialist in Endodontics / Researcher, Bezmialem Vakif University
Organization: Bezmialem Vakif University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20/5
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Asymptomatic Apical Periodontitis; Root Canal Infection; Periapical Diseases; Dental Pain
Keywords: EDDY Device; Sonic Irrigation; Root Canal Treatment; Apical Periodontitis; Postoperative Pain; Real-Time PCR; Randomized Controlled Trial
MeSH Terms: conditions — Periapical Diseases; Toothache; Periapical Periodontitis; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Parallel assignment of 40 participants into two groups: one receiving sonic irrigation using the EDDY device and the other receiving conventional syringe irrigation. Each participant received a single intervention without crossover.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EDDY Group (Experimental): Patients in this group received final irrigation using the EDDY sonic activation device after standard root canal instrumentation.
  Interventions: Device: EDDY Sonic Activation
- Conventional Irrigation Group (Active Comparator): Patients in this group received final irrigation with conventional syringe irrigation after standard root canal instrumentation.
  Interventions: Procedure: Conventional Syringe Irrigation

INTERVENTIONS:
Device: EDDY Sonic Activation — Sonic activation was performed using the EDDY device with 2.5% NaOCl and 17% EDTA solutions during final irrigation, following root canal preparation.
  Arms: EDDY Group
Procedure: Conventional Syringe Irrigation — Final irrigation was performed using syringe irrigation with 2.5% NaOCl and 17% EDTA solutions, without any activation.
  Arms: Conventional Irrigation Group

SUMMARY:
This randomized controlled clinical trial aimed to evaluate the effect of sonic activation using the EDDY device on root canal microbiota and postoperative pain in teeth with asymptomatic apical periodontitis. Forty patients were assigned to either a sonic activation group (EDDY) or a conventional irrigation group. Bacterial samples were collected before and after root canal treatment and analyzed using real-time PCR. Postoperative pain was assessed using a Numerical Rating Scale at various time intervals. The results showed that EDDY sonic activation significantly reduced bacterial load, while no statistically significant difference was found in postoperative pain between the groups.

DETAILED DESCRIPTION:
This prospective, randomized controlled clinical trial was conducted to assess the impact of sonic irrigation using the EDDY device on the reduction of intracanal microbiota and on postoperative pain following root canal treatment of teeth with asymptomatic apical periodontitis. Forty participants with single-rooted teeth were randomly allocated into two groups: the EDDY group, which received final irrigation activated with the EDDY sonic system, and the control group, which received conventional syringe irrigation. Microbiological samples were collected before and after instrumentation and were analyzed using real-time PCR to detect specific bacterial taxa. Postoperative pain levels were recorded using the Numerical Rating Scale at multiple time intervals up to 48 hours after treatment. The results demonstrated a statistically significant reduction in bacterial load in the EDDY group compared to the control group, but no significant difference in postoperative pain was observed. The findings support the use of EDDY sonic activation as an effective method for enhancing root canal disinfection.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* Presence of a single-rooted tooth diagnosed with asymptomatic apical periodontitis
* No previous endodontic treatment on the involved tooth
* Good general health (ASA I or II)
* Ability to provide informed consent

Exclusion Criteria:

* Teeth with internal or external resorption
* Pregnant or breastfeeding women
* Systemic antibiotic or anti-inflammatory drug use within the past 30 days
* Patients with periodontal pockets >4 mm on the affected tooth
* Known allergy to sodium hypochlorite or EDTA
* Patients who failed to attend postoperative pain follow-up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-20 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Change in Bacterial Load (CFU/mL) After Root Canal Treatment | Baseline and immediately after instrumentation (same visit)
  Bacterial samples were taken from the root canal before and after treatment. Quantitative changes in bacterial load were assessed using real-time PCR analysis of selected bacterial taxa.

SECONDARY OUTCOMES:
Postoperative Pain Level | 6, 12, 24, and 48 hours after treatment
  Postoperative Pain Level Patients were asked to rate their pain using the Numerical Rating Scale (range 0-10; 0 = no pain, 10 = worst possible pain) at 4 time points after treatment. Higher scores indicate greater pain intensity. Pain scores were compared between groups.
  [Time Frame: 6, 12, 24, and 48 hours after treatment]

CONTACTS AND LOCATIONS:
Overall Officials: Abdulkadir Tiftik, DDS, DDS, Principal Investigator — Bezmialem Vakif University, Faculty of Dentistry
Locations (1):
- Bezmialem Vakıf University, Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared because the study was conducted locally with a limited sample size, and there is no institutional plan or repository in place for data sharing.